CLINICAL TRIAL: NCT02721368
Title: Clinical Study of Neuramis® Volume Lidocaine to Evaluate the Efficacy and Safety for Temporary Restoring the Mid-face Volume
Brief Title: Neuramis® Volume Lidocaine Treatment in Patients With Loss of Mid-face Volume
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT_PRT_MVD01
Record Dates: First submitted 2016-03-14; First posted 2016-03-29 (Estimated); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational medical device (Experimental): Neuramis® Volume Lidocaine
  Interventions: Device: Neuramis® Volume Lidocaine
- Comparator medical device (Active Comparator): Juvederm® Voluma® with Lidocaine
  Interventions: Device: Juvederm® Voluma® with Lidocaine

INTERVENTIONS:
Device: Neuramis® Volume Lidocaine — hyaluronic acid filler
  Arms: Investigational medical device
Device: Juvederm® Voluma® with Lidocaine — hyaluronic acid filler
  Arms: Comparator medical device

SUMMARY:
The purpose of this study is to compare the safety and efficacy of Neuramis® Volume Lidocaine, which is a biomaterial prosthesis and graft, with Juvederm® Voluma® with Lidocaine, for the patients who need correction due to a moderate-to-severe volume loss in the mid-facial region by inducing temporary volume restoration in mid-facial region. After the pivotal study, extension study will be conducted to confirm long-term safety and efficacy.

DETAILED DESCRIPTION:
This is a multi-centered, randomized, double-blind, split-face clinical study on investigational device. The subjects in this clinical trial receive application of the investigational device on the right and left side of the mid-facial region (Neuramis® Volume Lidocaine or Juvederm® Voluma® with Lidocaine). After the pivotal study, extension study will be conducted to confirm long-term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Subject aged between 35 and 65.
2. Mid-facial region symmetrical, severity greater than MFVDS moderate-to-severe level

Exclusion Criteria:

1. Those who have anticoagulant therapy, antiplatelet therapy, and non-steroidal anti-inflammatory drugs
2. Those who have history of receiving the procedures which are considered to affect on the assessment of this clinical trial.
3. Those who has thin skin in the mid-facial area
4. Those with hypersensitivity to sodium hyaluronate or lidocaine or amide type local anesthetics

<Extension Study>

Inclusion Criteria:

1. Participated in the pivotal study and completed the end of study visit
2. Agreed not to receive any procedure or treatment that may have an effect on the restoration of the mid-face volume while participating in the extension study

Exclusion Criteria

1. Those who have following procedual history between completion of the pivotal study and entry of extension study

   - facial plastic surgery, tissue grafting or tissue augmentation using implant, thread lifting
2. Subjects with asymmetric MVD(Mid-face volume deficit) or facial scar interfering with accurate assessment

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
Ratio of subjects defined as improved by independent photograph evaluator according to the overall Mid-Face Volume Deficit Scale(MFVDS) | 24 weeks
  MFVDS 0- None, 1-Minimal, 2-Mild, 3-Moderate, 4-Significant, 5-Severe The lower score, the better condition.
Ratio of subjects defined as improved by independent photograph evaluator according to the overall Mid-Face Volume Deficit Scale(MFVDS) | 104 weeks
  Primary outcome for extension study

SECONDARY OUTCOMES:
The changes in overall Mid-Face Volume Deficit Scale(MFVDS) at each visit | 104 weeks
Ratio of subjects defined as improved by blinded investigators and the subjects according to the Global Aesthetic Improvement Scale (GAIS) | 104 weeks

CONTACTS AND LOCATIONS:
Overall Officials: BeomJoon Kim, Principal Investigator — Chung-Ang Univ. Medical Center
Locations (1):
- Chung-Ang Univ. Medical Center, Seoul, Dongjak-gu, South Korea

IPD SHARING:
Plan to Share IPD: Undecided